CLINICAL TRIAL: NCT05771753
Title: Comparison of Core Stabilization and Dynamic Stretching Exercises on Symptoms Severity and Quality of Life in Primary Dysmenorrhea
Brief Title: Comparison of Core Stabilization and Dynamic Stretching Exercises in Primary Dysmenorrhea
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/22/0548
Record Dates: First submitted 2023-02-28; First posted 2023-03-16 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2023-03

CONDITIONS: Primary Dysmenorrhea
MeSH Terms: interventions — Muscle Stretching Exercises

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stretching Exercises (Experimental): 6 stretching exercise for 8 weeks
  Interventions: Other: Stretching Exercises
- Dynamic core stabilizing exercises (Experimental): 6 strengthening exercises for 8 weeks
  Interventions: Other: Dynamic core stabilizing exercises

INTERVENTIONS:
Other: Stretching Exercises — 6 stretching exercises 2 repetitions x1 set, 3 days/week and targeted muscles stretching (Lower Back, Lower limb)
  Arms: Stretching Exercises
Other: Dynamic core stabilizing exercises — This group received core stabilizing exercises 2 repetitions x1 set, 3 days/week and the targeted muscles were abdominals, lower back, and lower limb.
  Arms: Dynamic core stabilizing exercises

SUMMARY:
A randomize control study will be conducted, in which data will be collected from young girls having primary dysmenorrhea with the calculated sample size of 17 in each group, questionnaire will be provided to collect the data and then according to sample size number the participants will be randomly assign to the group A and B. group A will perform stretching exercises for eight weeks and group B will perform core stabilizing exercises for 8 weeks, pre and post readings before starting exercises and after eight weeks will be taken. Four different types of tools will be used, for primary dysmenorrhea WALIDD scale will be used, to measure the pain intensity, frequency, duration and severity the PFSD scale will be used and for measuring the strength the side bridge test will be used and to check the effects of primary dysmenorrhea on quality of life, McGill quality of life questionnaire will be used. This study will provide the information that which exercises i-e stretching or strengthening are more effective in reducing the intensity, frequency, duration and severity of pain in primary dysmenorrhea.

DETAILED DESCRIPTION:
Primary dysmenorrhea is a Greek term which means difficult flow and the term describe painful periods. The pain is usually felt in the lower abdomen but sometimes it may radiate in thighs and to the back. Primary dysmenorrhea is the most common type of gynecological disorder among females worldwide. Some females may feel some associated symptoms like nausea, vomiting diarrhea, headache, dizziness and in severe conditions syncope. All of these symptoms occur usually in females with normal pelvic anatomy and symptoms occur just before menses. Primary dysmenorrhea occurs 6-12 months after the onset of ovulation cycle. Primary dysmenorrhea can be distinguished from secondary dysmenorrhea on the basis of symptoms and other pelvic or reproductive organ disorders. Endometriosis is the most common cause of secondary dysmenorrhea, in secondary dysmenorrhea pain starts few days before the onset of menstrual cycles and may last longer than the cycle. The chances of secondary dysmenorrhea are more prevalent in females above the age of 20. A complete pelvic examination should be performed in females who are sexually active and have dysmenorrhea and those who are suspected to have endometriosis. In general population the prevalence of Primary dysmenorrhea is about 47-80%. Seventy five to eighty five percent of female have said to report that the symptoms of primary dysmenorrhea are mild. Primary dysmenorrhea is not life threatening and does not cause any disabilities but some researches have said that most young girls are reported to be absent from school/college and not being able to perform any activity due to the severity of pain. Some evidence shows the link between dysmenorrhea and prostaglandin, the level of prostaglandin is said to be increased and leads to uterine contraction and ischemia. The release of prostaglandin leads to excessive uterine contraction and the constriction of small endometrial blood vessels leads to ischemia and thus pain. The level of prostaglandin is said to be increased during premenstrual phase in which progesterone level decreases and the level of prostaglandin increases in endometrial cells by the action of membrane phospholipids. The action of prostaglandin synthesis inhibitors plays an important role in pain relief. Another interesting factor shows the link between physical activity and dysmenorrhea.

Females who perform physical activities like exercise for the purpose of developing or maintaining fitness have reported to be going through less pain and behavioral changes.

Physical activities and exercises are believed to have reduced the level of stress and stress related symptoms. When we do exercise endorphins hormones are released from brain which increases the pain threshold and have said to improve the mood of the person performing exercise. It has also been observed that performing isometric exercises for 8 weeks has reduced the intensity and duration of pain but has no effects on the amount of bleeding. Performing stretching exercises for 8 weeks has also reduced the severity and length of pain in young girls and they have reported to be taking less medicine. The purpose of this research is to provide the information that which exercises i-e stretching or strengthening are more effective in reducing the intensity, frequency, duration and severity of pain in primary dysmenorrhea.

ELIGIBILITY:
Inclusion Criteria:

* Unmarried young girls of age 18-25.
* Nulliparous women
* Voluntarily wants to participate

Exclusion Criteria:

* Female with History of any specific disease
* Having symptoms such as tingling sensation
* Any history of regular physical activity 3days/week [daily average 30-45 minutes] were ruled out of the study.

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-04-25 (Estimated); Study Completion 2023-04-25 (Estimated)

PRIMARY OUTCOMES:
WaLIDD (working ability, Location, Intensity, Days of pain, Dysmenorrhea) score | 8 weeks
  A scale type survey incorporating features of primary dysmenorrhea Score: 0 without dysmenorrhea, I-4 mild dysmenorrhea, 5-7 moderate dysmenorrhea, 8-12 severe dysmenorrhea.
side bridge test | 8 weeks
  side bridge test is use to check the strength of individuals
McGill Quality of life | 8 weeks
  A questionnaire used to check the effects of diseases on the quality of life
PFSD (pain, frequency, severity, duration) scale | 8 weeks
  A self reported pain questionnaire that captures the multidimensionality of pain A composite score was derived by multiplying the number of days of pain, the level of usual pain, and the level of worst pain and then dividing the product by 10.

CONTACTS AND LOCATIONS:
Overall Officials: Iqra Abdul Ghafoor, ppdpt, Principal Investigator — Riphah International University
Locations (1):
- University of Sialkot, Sialkot, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Iacovides S, Avidon I, Baker FC. What we know about primary dysmenorrhea today: a critical review. Hum Reprod Update. 2015 Nov-Dec;21(6):762-78. doi: 10.1093/humupd/dmv039. Epub 2015 Sep 7. PMID 26346058
- [Background] Karout S, Soubra L, Rahme D, Karout L, Khojah HMJ, Itani R. Prevalence, risk factors, and management practices of primary dysmenorrhea among young females. BMC Womens Health. 2021 Nov 8;21(1):392. doi: 10.1186/s12905-021-01532-w. PMID 34749716
- [Background] Bernardi M, Lazzeri L, Perelli F, Reis FM, Petraglia F. Dysmenorrhea and related disorders. F1000Res. 2017 Sep 5;6:1645. doi: 10.12688/f1000research.11682.1. eCollection 2017. PMID 28944048
- [Background] De Sanctis V, Soliman A, Bernasconi S, Bianchin L, Bona G, Bozzola M, Buzi F, De Sanctis C, Tonini G, Rigon F, Perissinotto E. Primary Dysmenorrhea in Adolescents: Prevalence, Impact and Recent Knowledge. Pediatr Endocrinol Rev. 2015 Dec;13(2):512-20. PMID 26841639
- [Background] Brawn J, Morotti M, Zondervan KT, Becker CM, Vincent K. Central changes associated with chronic pelvic pain and endometriosis. Hum Reprod Update. 2014 Sep-Oct;20(5):737-47. doi: 10.1093/humupd/dmu025. Epub 2014 Jun 11. PMID 24920437
- [Background] Lindh I, Ellstrom AA, Milsom I. The effect of combined oral contraceptives and age on dysmenorrhoea: an epidemiological study. Hum Reprod. 2012 Mar;27(3):676-82. doi: 10.1093/humrep/der417. Epub 2012 Jan 17. PMID 22252090
- [Background] Guimaraes I, Povoa AM. Primary Dysmenorrhea: Assessment and Treatment. Rev Bras Ginecol Obstet. 2020 Aug;42(8):501-507. doi: 10.1055/s-0040-1712131. Epub 2020 Jun 19. PMID 32559803